CLINICAL TRIAL: NCT03728686
Title: The Hemodynamic Response to Endotracheal Intubation at Different Time of Fentanyl Given During Induction: a Randomized Controlled Trial
Brief Title: Response to Endotracheal Tube Intubation at Different Time of Fentanyl Given During Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chien-Chung,Huang (Other)
Responsible Party: Sponsor-Investigator, Chien-Chung,Huang, attending physician, department of anesthesiology, Mackay Memorial Hospital
Organization: Mackay Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 16MMHIS097e
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Intubation, Intratracheal
Keywords: Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3mins (Experimental): Different given time: Fentanyl 2mcg/kg was given at either time 3 minutes before intubation
  Interventions: Other: Different given time
- 2mins (Active Comparator): Different given time: Fentanyl 2mcg/kg was given at either time 2 minutes before intubation
  Interventions: Other: Different given time
- control (No Intervention): Different given time: Fentanyl 2mcg/kg was given at either time 1 minute before intubation

INTERVENTIONS:
Other: Different given time — Fentanyl 2mcg/kg (F) was given at either 1,2,3 minutes before intubation
  Arms: 2mins; 3mins

SUMMARY:
Opioids have been used to modify the hemodynamic response associated with laryngoscopy and tracheal intubation. To seek the correlation of Fentanyl given time, we will analysis the data collected from vital signs monitoring machine. Patients'details will be recorded too.

DETAILED DESCRIPTION:
Laryngoscopy and intubation often provoke hypertension and tachycardia due to the stimulation both sympathetic and sympathoadrenal activities. While the adverse hemodynamic effects of laryngoscopy and endotracheal intubation can precipitate myocardial ischemia, even in patients without hypertension, the responses are exaggerated in patients with hypertension . In the previous studies , many drugs, including opioids and beta-blockers, have been used to modify the hemodynamic response associated with laryngoscopy and tracheal intubation. To seek the correlation of Fentanyl given time, we will analysis the data collected from vital signs monitoring machine.

All patients were premedicated with Midazolam 0.1mg/kg , Lidocaine 0.5mg/kg (L), Propofol 2mg/kg (P), Rocuronium 1mg/kg (R) before induction of general anesthesia. Laryngoscopy lasting a maximum of 30 s was attempted 3 min after administration of the induction agents. Fentanyl 2mcg/kg was given at different time before intubation.

ELIGIBILITY:
Inclusion Criteria:

* with American Society of Anesthesiologists (ASA) physical status classification 1&2
* undergo elective surgery
* intubation

Exclusion Criteria:

* Opioids allergy history

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
heart rate | 0-10 minutes during induction
  heart rate
systolic blood pressure | 0-10 minutes during induction
  systolic blood pressure
diastolic blood pressure | 0-10 minutes during induction
  diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Chicn-Chung Huang, MD, Study Director — Mackay Memorial Hospital
Locations (1):
- MacKay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parida S, Ashraf NC, Mathew JS, Mishra SK, Badhe AS. Attenuation of the haemodynamic responses to tracheal intubation with gabapentin, fentanyl and a combination of both: A randomised controlled trial. Indian J Anaesth. 2015 May;59(5):306-11. doi: 10.4103/0019-5049.156885. PMID 26019356
- [Background] Sawano Y, Miyazaki M, Shimada H, Kadoi Y. Optimal fentanyl dosage for attenuating systemic hemodynamic changes, hormone release and cardiac output changes during the induction of anesthesia in patients with and without hypertension: a prospective, randomized, double-blinded study. J Anesth. 2013 Aug;27(4):505-11. doi: 10.1007/s00540-012-1552-x. Epub 2013 Jan 12. PMID 23314694
- [Background] Derbyshire DR, Chmielewski A, Fell D, Vater M, Achola K, Smith G. Plasma catecholamine responses to tracheal intubation. Br J Anaesth. 1983 Sep;55(9):855-60. doi: 10.1093/bja/55.9.855. PMID 6615672
- [Background] Shribman AJ, Smith G, Achola KJ. Cardiovascular and catecholamine responses to laryngoscopy with and without tracheal intubation. Br J Anaesth. 1987 Mar;59(3):295-9. doi: 10.1093/bja/59.3.295. PMID 3828177
- [Background] Martin DE, Rosenberg H, Aukburg SJ, Bartkowski RR, Edwards MW Jr, Greenhow DE, Klineberg PL. Low-dose fentanyl blunts circulatory responses to tracheal intubation. Anesth Analg. 1982 Aug;61(8):680-4. PMID 7201271